CLINICAL TRIAL: NCT06951672
Title: The AMEND TS Early Feasibility Study is a Prospective, Single-arm, Multi-center Study to Evaluate the Safety and Function of the AMEND(TM) Trans-Septal System for MR Reduction; Up to 15 Subjects Will be Enrolled in up to 7 Investigational Centers in the U.S. and Canada With a 30d Safety Endpoint
Brief Title: AMEND TS Early Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valcare Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP - 0001762
Record Dates: First submitted 2025-04-04; First posted 2025-04-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Functional MR 3 or Greater
Keywords: MR reduction; mitral regurgitation; Heart valve; annuloplasty ring; functional mitral regurgitation; mitral valve
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- prospective, single arm, open trial to evaluate the safety, functionality of the AMEND TS System (Experimental): The AMEND TS EFS is a prospective, single arm, open clinical trial designed to evaluate the safety and functionality of the AMENDTM Trans-Septal System for MR reduction in patients suffering from functional mitral regurgitation.
  This study will evaluate the safety and functionality of the AMEND™ Trans-Septal System for annuloplasty as a therapy for mitral regurgitation.
  Interventions: Device: This study will evaluate the safety and functionality of the AMEND™ Trans-Septal System for annuloplasty as a therapy for mitral regurgitation.

INTERVENTIONS:
Device: This study will evaluate the safety and functionality of the AMEND™ Trans-Septal System for annuloplasty as a therapy for mitral regurgitation. — The ability to deploy the annuloplasty ring in a percutaneous fashion affords an improved safety profile for surgical candidates, as well as surgical style solution for those patients that are at elevated risk for surgery due to comorbidities and advanced age. This early feasibility study allows treatment of higher risk surgical candidates with a surgical- level annuloplasty repair therapy by the AMEND™ Implant.

SUMMARY:
Valcare Medical AMEND Trans-Septal System is a mitral valve repair annuloplasty ring implanted in a trans-catheter method intended for correction of mitral regurgitation. It is designed to be used as standalone therapy or in combination with other repair treatments.

DETAILED DESCRIPTION:
Objective: The purpose of this clinical investigation, the AMEND TS Early Feasibility Study, is to evaluate the safety and functionality of the AMEND Trans-Septal System for annuloplasty as treatment of mitral regurgitation.

Device Description: The AMENDTM Trans-Septal System consists of a semi-rigid annuloplasty ring (implant), a delivery system (catheter), and accessories (Stage, Introducer sheath). The device is delivered through a catheter using a trans-septal approach and implanted in the beating heart on the atrial surface of the mitral valve annulus similar to surgical annuloplasty rings.

Indications for Use: The device is indicated to treat patients with mitral regurgitation using a percutaneous direct annuloplasty approach

Number of subjects and sites: Up to fifteen (15) subjects will be enrolled to the study procedure in up to 7 investigational centers in the U.S. and Canada

Study Population: Subjects with symptomatic moderate-to-severe (3+) or severe (4+) functional mitral regurgitation that is anatomically amenable to transcatheter mitral annuloplasty.

Study Duration: 5 years

ELIGIBILITY:
Inclusion Criteria:

1. Patient age >21
2. The patient will benefit from isolated mitral valve annuloplasty for mitral regurgitation without the need for concomitant cardiovascular surgical procedures such as coronary artery bypass or another valve reconstruction or replacement
3. Symptomatic functional MR≥3+
4. NYHA functional capacity ≥2
5. LV Ejection Fraction > 30%, LVEDD < 68 mm
6. The subject meets the anatomical eligibility criteria for available implant size(s)
7. The subject is at high risk for mitral valve surgery as assessed by the center's heart team for mitral procedures.
8. The subject has been stable and on a stable pharmacological regimen for heart failure for at least 1 month prior to inclusion
9. Femoral vein access and transseptal device access is determined to be feasible by the implanting investigator
10. The patient is willing to comply with study procedures and is available to return to the implant center for follow-up visits
11. Informed consent documentation signed and dated confirming that the patient has been adequately informed of all aspects related to his/her participation in the clinical study and is willing to participate.

Exclusion Criteria:

1. The patient has mitral incompetence where an annuloplasty ring will not contribute to its repair
2. Cardiac or non-cardiac major or progressive disease, which in the investigator's discretion produces an unacceptable increased risk to the patient.
3. Life expectancy of less than 12 months
4. The subject is non-operable and is not eligible for TEER, to allow bailout
5. Heavily calcified mitral annulus or leaflets
6. Previous or active endocarditis.
7. Active infection
8. A previously implanted prosthetic aortic valve or mitral intervention
9. Cardiovascular intervention within 30 days prior to study procedure
10. GFR <30 ml/min
11. The patient has had an ischemic coronary event within 30 days prior to study procedure
12. The patient has clinically significant coronary artery disease requiring re- vascularization
13. The subject is contraindicated to general anesthesia
14. The subject is unable to take anti-platelet or anti-coagulant medications
15. A known allergy to nickel
16. Severe allergy to contrast media
17. Significant right ventricle dysfunction
18. Left atrial thrombus
19. A cerebral vascular event (CVA or TIA) within the past 12 months
20. A mitral valve anatomy which may preclude proper AMEND™ treatment
21. Pulmonary systolic hypertension (estimated SPAP > 70 mmHg at rest), determined by echocardiography
22. Pregnant (for women in the reproductive age, blood HCG test result positive) or lactating patient
23. Drug or alcohol abuse
24. Participation in concomitant research studies of investigational products
25. Any planned cardiac surgery or interventions within the next 7 months
26. Implant or revision of any rhythm management device (cardiac resynchronization therapy (CRT) or cardiac resynchronization therapy device (CRT-D)) or implantable cardioverter defibrillator within the prior month
27. Hypotension (systolic pressure <90 mm Hg) or requirement for inotropic support or mechanical hemodynamic support
28. Status 1 heart transplantation or prior orthotopic heart transplantation
29. Subjects in whom transesophageal echocardiography is contraindicated or high risk

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint: Composite of death (all-cause), stroke, myocardial infarction (MI), or non-elective cardiovascular surgery for device related complications at 30 days. | 30 days
  The definitions of the SAEs are based on the recommendation of the Mitral Valve Academic Research Consortium (MVARC) (Stone, 2015).

SECONDARY OUTCOMES:
Secondary Endpoint: Performance Endpoint | 30 days
  Technical success of ring delivery, implantation and delivery system retrieval determined at the end of implantation procedure based on the following:
  * Absence of procedural mortality
  * Freedom from emergency surgery or corrective treatment related to the device or access procedure
  * Successful access, delivery to the LA, and retrieval of the delivery system
  * Correct positioning of the implant evaluated by echocardiography after procedure completion
  * Adequate implant quadrant fixation evaluated by echocardiography after procedure completion

OTHER OUTCOMES:
Additional Endpoints | 6 months and 1 year
  Safety at 6 months; a composite of all-cause death, stroke, MI, or non-elective cardiovascular surgery for device related complications

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Meerkin, CMO, MD, Study Director — Valcare Medical
Locations (11):
- United States (11):
  - Banner University Medical Center - Phoenix, Phoenix, Arizona
  - Scripps Health, La Jolla, California
  - Piedmont Healthcare, Atlanta, Georgia
  - Ascension St. Vincent, Indianapolis, Indiana
  - Columbia University Medical Center (CUMC), New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Saint Thomas Research Institute, Nashville, Tennessee
  - University of Texas Health Science Center (UTH), Houston, Texas
  - Methodist Hospital HCA, San Antonio, Texas
  - Intermountain Health, Murray, Utah

IPD SHARING:
Plan to Share IPD: Undecided